CLINICAL TRIAL: NCT01649973
Title: Study for Appropriate Operating Table Height for Endotracheal Intubation Under Direct Laryngoscopy
Status: Completed | Type: Observational
Sponsor: National Medical Center, Seoul (Other)
Responsible Party: Principal Investigator, Mi Ja Yun, MD, PhD, Professor, National Medical Center, Seoul
Other Study IDs: SeoulNUBH-B-1003-096-012
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Larynx
MeSH Terms: conditions — Laryngeal Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Laryngeal view of the patient and anesthesiologist's discomfort level during endotracheal intubation in relation to the various heights of operating table has not been investigated. The investigators hypothesis is higher table height will improve the laryngeal exposure.

DETAILED DESCRIPTION:
Eight anesthesiologists will be participated. For each anesthesiologist, 20 patients will be enrolled and they will be randomly allocated into one of 4 groups; T10, T8, T6 or T4. The height of operating table will be adjusted prior to commencement of anesthesia induction to place the patient's forehead at one of four anesthesiologist's dermatome levels (T10, T8, T6 or T4) depending on the group. The best laryngeal views will be graded before and after the anesthesiologist's postural change to improve laryngeal visualization of the patient during intubation. Subjective and objective measurement of anesthesiologists' joint flexion during intubation and discomfort ratings for the mask ventilation or intubation will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* have experiences of more than 100 cases of endotracheal intubation

Exclusion Criteria:

* have acute or chronic musculoskeletal disease or pain

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: certificated anesthesiologists
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
larynx | larynx

CONTACTS AND LOCATIONS:
Overall Officials: Mija Yun, Study Chair — National Medical Center, Seoul

REFERENCES:
- [Derived] Lee HC, Yun MJ, Hwang JW, Na HS, Kim DH, Park JY. Higher operating tables provide better laryngeal views for tracheal intubation. Br J Anaesth. 2014 Apr;112(4):749-55. doi: 10.1093/bja/aet428. Epub 2013 Dec 18. PMID 24355831